CLINICAL TRIAL: NCT00504075
Title: A Phase III, Multicenter, Open-Label Study To Evaluate the Efficacy and Safety of GAMMAPLEX® in Chronic Idiopathic Thrombocytopenic Purpura
Brief Title: A Study to Find How Safe and Effective GAMMAPLEX® is in Subjects With Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMX02
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Results first posted 2012-06-06 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic Thrombocytopenic Purpura; Bleeding disorders; Immune System and Disorders
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Hemostatic Disorders; Immune System Diseases | interventions — gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gammaplex (intravenous immunoglobulin) (Experimental)
  Interventions: Biological: Gammaplex, intravenous immunoglobulin

INTERVENTIONS:
Biological: Gammaplex, intravenous immunoglobulin — Dosage form: Gammaplex® is a sterile liquid of 5 % w/v normal immunoglobulin. Gammaplex® contains 5 g/100 mL of human normal immunoglobulin (i.e. 50 g/L, of which virtually 100% is IgG).
  The first course of GAMMAPLEX will be administered as an intravenous infusion of 1 g/kg on each of 2 consecutive days. If required, a further 1 or 2 courses on the same dosage regimen may be administered in the period Day 32 to Day 90 following the first course of GAMMAPLEX.
  Other Names: Gammaplex

SUMMARY:
To determine if GAMMAPLEX raises the platelet count of subjects with chronic ITP to a threshold of 50 x 109/L, similar to that of published response >60%. Also to assess the safety of GAMMAPLEX and determine if platelet counts are maintained at 50 x 109/L in subjects with chronic ITP for.

DETAILED DESCRIPTION:
The primary objective is to determine if BPL's GAMMAPLEX raises the platelet count of subjects with chronic ITP to a threshold of 50 x 109/L, similar to that of published response >60%. The secondary objectives are: 1) to determine the safety of GAMMAPLEX at the dosage used in this study. 2) to determine if GAMMAPLEX maintains platelet counts of ³ 50 x 109/L in subjects with chronic ITP for a period of time similar to that of a published data.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged between 18 and 70 years.
2. Confirmed diagnosis of chronic ITP of at least 6 months duration.
3. Platelet count of less than or equal to 20 x 10 9/L at enrollment.
4. Absence of other conditions that, in the opinion of the investigator, could cause thrombocytopenia.
5. If subjects were treated with corticosteroids the treatment regimen/dose must have been stable (for a minimum of 2 weeks before screening). The dose of corticosteriod or other immunosuppressant should have remained constant until Day 32. 6) If subjects were being treated with cyclophosphamide, azathioprine or attenuated androgens, the treatment regimen and dose must have been stable for a minimum of 2 months before Day 1. The dose of corticosteriod or other immunosuppressant should have remained constant until Day 32. 7) Splenectomized subjects and both Rh(D)+ and Rh(D)- subjects may be included.

8) The subject has signed an informed consent form (subjects must be at least 18 years old), and/or the subject's legal guardian has signed the informed consent form if indicated 9) If a subject is a female of child-bearing potential, she must have a negative result on a urine-based HCG pregnancy test.

10) If a subject is a female who is or becomes sexually active, she must practice contraception by using a method of proven reliability for the duration of the study.

Exclusion Criteria:

1. A history of any severe or anaphylactic reaction to blood or any blood-derived product, or any severe reaction to IGIV or any other IgG preparation.
2. Intolerance to any component of the investigational product.
3. Received any live virus vaccine within the last 3 months prior to Day1.
4. Received an IGIV preparation within 1 month prior to Day 1.
5. Were currently receiving, or has received, any investigational agent within the 1 month prior to Day 1.
6. Received any blood, blood product, or blood derivative within the 1 month prior to Day 1.
7. Received Rituximab within the 3 months before Day 1.
8. Pregnant or nursing.
9. Tested positive for any of the following at screening: HBsAg, NAT for HCV, NAT for HIV, Antibodies to HCV or HIV 1 or 2.
10. Had levels greater than 2.5 times the upper limit of normal at screening, as defined by the central laboratory, of alanine aminotransferase or aspartate aminotransferase.
11. Had severe renal impairment (defined as serum creatinine greater than 2 times the upper limit of normal or BUN greater than 2.5 times the upper limit of normal for the range of the laboratory doing the analysis); on dialysis; a history of acute renal failure.
12. Known to have abused alcohol, opiates, psychotropic agents, or other chemicals or drugs within the past 12 months.
13. History of deep vein thrombosis (DVT) or thrombotic complications of IGIV therapy.
14. Any history or sign of hyperviscosity, transient ischemic attack (TIA), stroke, other thromboembolic event, or unstable angina.
15. Suffered from any acute or chronic medical conditions (e.g., renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing enteropathy) that, in the opinion of the investigator, may interfere with the conduct of the study.
16. An acquired medical condition, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (defined as an absolute neutrophil count (ANC) < 1 x 109/L).
17. Non-controlled arterial hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg).
18. Anemic (hemoglobin <10 g/dL) at screening.
19. Unlikely to adhere to the protocol requirements of the study or is likely to be uncooperative.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Aldwinckle, MD, Principal Investigator — Bio Products Laboratory
Locations (30):
- United States (7):
  - Mid Florida Hematology & Oncology, Orange City, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - New York Hospital / Cornell University, Division of Pediatrics, New York, New York
  - Department of Pediatrics, SUNY at Stony Brook, Stony Brook, New York
  - Oregon Health & Science University, Portland, Oregon
  - Cancer Care Centers of South Texas, San Antonio, Texas
- Argentina (9):
  - Hospital Churruca, Capital Federal, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - CER San Juan, San Juan, San Juan Province
  - Instituto de Diagnóstico Hematológico Ambulatorio (IDHEA), Rosario, Sante Fe
  - I. A. D. T. (Instituto Argentino de Diagnóstico y Tratamiento), Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clinicas Dr. Norberto Quirno (CEMIC), Buenos Aires
  - J.R. Vidal Hospital, Corrientes
  - Hospital Privado de Cordoba, Córdoba
- India (14):
  - Apollo Hospitals, Hyderabad, Andhra Pradesh
  - Mahavir Hospital, Hyderabad, Andhra Pradesh
  - City Cancer Centre,, Suryarao Pet, Vijayawada, Andhra Pradesh
  - M. S Ramaiah Hospital, Karnataka, Bangalore
  - Vedanta, Ahmedabad, Gujarat
  - Gurukrupa Hospital, Ahmedabad, Gujarat
  - M S Patel Cancer Centre, Shree Krishna Hospital, Gokal Nagar, Karamsad, Gujarat
  - Manipal Hospital, Bangalore, Karnataka
  - Vinaya Hospital & research Centre, Mangalore, Karnataka
  - Kasturba Medical College, Manipal Acunova KMC Research Centre, Mangalore, Karnataka
  - Father Muller Medical College Hospital, Mangalore, Karnataka
  - Deenanath Mangeshkar Hospital, Pune, Maharashtra
  - S.K. Soni Hospital Sect 5, Jaipur, Rajasthan
  - Sir Ganga Ram Hospital, New Delhi

REFERENCES:
- [Derived] Dash CH, Gillanders KR, Stratford Bobbitt ME, Gascoigne EW, Leach SJ. Safety and efficacy of Gammaplex(R) in idiopathic thrombocytopenic purpura (ClinicalTrials.gov--NCT00504075). PLoS One. 2014 Jun 3;9(6):e96600. doi: 10.1371/journal.pone.0096600. eCollection 2014. PMID 24892422
- See also: Sponsor website — http://www.bpl.co.uk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First enrollment: 04 September 2007. Last Subject completed: 05 August 2011. Thirty-five sites in the United States, India and Argentina, all hospital clinics.
Pre-assignment Details: This was an open label study. All enrolled subjects received study medication.
Groups:
- GAMMAPLEX: The first course of GAMMAPLEX was administered as an intravenous infusion of 1g/kg on each of 2 consecutive days. If required, a further 1 or 2 courses on the same dosage regimen was administered in the period Day 32 to Day 90 following the first course of GAMMAPLEX.
Period: Overall Study
Arm/Group | GAMMAPLEX
Started | 35
Completed | 27
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1
Not completed — Required other therapeutic intervention | 1

BASELINE CHARACTERISTICS:
Arm/Group | GAMMAPLEX
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 29
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 9
  Argentina | 5
  India | 21

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Chronic ITP Treated With Gammaplex Whose Platelet Count Reached a Threshold of 50 x 10^9/L.
Description: The number of subjects with chronic ITP treated following treatment with Gammaplex who attained a platelet count of ≥ 50 x 10^9/L by Day 9.
Time Frame: 9 days
Population: Any subject who started treatment with GAMMAPLEX and whose central laboratory results taken prior to infusion on Day 1 were within specified protocol parameters, was included in the intent-to-treat (ITT) population for analysis of efficacy and safety.
Measure: Number; unit: participants
Arm/Group | GAMMAPLEX
Number analyzed (Participants) | 35
participants | 29 [60 to 100]

2. Secondary Outcome: The Safety of GAMMAPLEX at the Dosage Used in This Study.
Description: The safety variables used to assess safety were the following:
  * Adverse events
    * The number and percent of infusions with at least 1 adverse event(AE) that occurs during an infusion or within 72 hours after the infusion stops
    * Nature, severity, and frequency of AEs
    * Suspected unexpected serious adverse reactions (SUSARs)
  * Vital signs
  * Clinical laboratory tests and Direct Coombs' Test
  * Transmission of viruses
  * Physical examination
Time Frame: AEs were documented from the date the informed consent form was signed until the End of Study visit on Day 90.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects with product related SAEs
Arm/Group | GAMMAPLEX
Number analyzed (Participants) | 35
% of subjects with product related SAEs | 8.6 [1.8 to 23.1]

3. Secondary Outcome: Duration of Time That the Platelet Count of Subjects With Chronic ITP Treated With Gammaplex Remained ≥ 50 x 10^9/L.
Description: Blood samples were collected to measure platelet counts and the duration of time for which the platelet count remained ≥50 x 10^9/L was measured.
Time Frame: Days 1, 2, 3, 5, 9, 14, 21, 32.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | GAMMAPLEX
Number analyzed (Participants) | 35
days | 10 [7 to 14]

ADVERSE EVENTS:
Time Frame: An event was only included in the analysis of Adverse Events (AEs) if it had an onset date between the first GAMMAPLEX infusion and 30 days after the last GAMMAPLEX infusion, inclusive.
Arm/Group | GAMMAPLEX
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 21/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAMMAPLEX (N=35)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAMMAPLEX (N=35)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (3)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 4 (7)
Hypertension (Vascular disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (General disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 7 (7)
Pyrexia (General disorders) | 6 (10)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (11)
Headache (Nervous system disorders) | 11 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the Study results will be allowed only with prior written approval from Sponsor, said consent not to be unreasonably withheld. At the request of Sponsor, the Institution and/or Investigator shall delete any Confidential Information pertaining to Sponsor's Inventions from any proposed publications prior to submitting or presenting the materials. Any and all publications will give appropriate recognition of any support received from Sponsor.